CLINICAL TRIAL: NCT00184444
Title: Effect of Increased Oxygenation in the Air During Endurance Training in Stable Angina Pectoris Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 094-2004
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Angina Pectoris
Keywords: angina pectoris; hyperoxia; endurance training; stroke volume; cardiac perfusion
MeSH Terms: conditions — Angina Pectoris; Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxic Interval training (Experimental): 4 x 4 minutes interval training with 100% oxygenated air
  Interventions: Behavioral: Hypoxic interval training
- Normoxic interval training (Experimental): 4 x 4 minutes interval training in normoxic air
  Interventions: Behavioral: Normoxic interval training

INTERVENTIONS:
Behavioral: Hypoxic interval training — 4 x 4 minutes interval training in hypoxic air, 3 times per week at 90-95% HR max
  Arms: Hypoxic Interval training
Behavioral: Normoxic interval training — 4 x 4 minutes normoxic interval training, 3 times per week at 90-95% HR max
  Arms: Normoxic interval training

SUMMARY:
The study investigates whether endurance training breathing 100% oxygen gives a additional improvement of maximal oxygen uptake in stable Angina Pectoris patients, compared to training without extra oxygen supplementation. In addition work economy, stroke volume and cardiac perfusion is measured.

The hypothesis of the study is that increased oxygenation of the air increases performance, stroke volume, work economy and cardiac perfusion.

ELIGIBILITY:
Inclusion Criteria:

* stable angina pectoris age 18-75

Exclusion Criteria:

* unstable angina pectoris
* Limitations to exercise other than coronary artery disease
* Participants in other study interventions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake | Baseline and post training

SECONDARY OUTCOMES:
Cardiac perfusion | Baseline and post training
work economy | Baseline and post training
cardiac output | baseline and post training

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Støylen, MD, Study Director — Norwegian university of sience and technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Karlsen T, Hoff J, Stoylen A, Skovholdt MC, Gulbrandsen Aarhus K, Helgerud J. Aerobic interval training improves VO2 peak in coronary artery disease patients; no additional effect from hyperoxia. Scand Cardiovasc J. 2008 Oct;42(5):303-9. doi: 10.1080/14017430802032723. PMID 18609057